CLINICAL TRIAL: NCT04517227
Title: A Single-Arm Open-Label Pilot Study of Combination Therapy of TACE and Ablation With Durvalumab in A Selected Hepatocellular Carcinoma Population at Intermediate Stage
Brief Title: The Combination Therapy of TACE and Ablation With Durvalumab in Hepatocellular Carcinoma at Intermediate Stage (TAD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zheng-Gang Ren, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-19-20285
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): All patients enrolled with receive the sequential therapy of TACE, ablation and durvalumab.
  Interventions: Drug: Durvalumab; Procedure: Transcatheter Hepatic Arterial Chemoembolization (TACE); Procedure: Ablation

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is a human monoclonal antibody (mAb) of the immunoglobulin G (IgG) 1 kappa subclass that inhibits binding of PD-L1 and is being developed by AstraZeneca/MedImmune for use in the treatment of cancer.
  Other Names: IMFINZI
Procedure: Transcatheter Hepatic Arterial Chemoembolization (TACE) — TACE techniques have been described in the NCCN and ESMO-ESDO guidelines, including cTACE and DEB-TACE.
Procedure: Ablation — In this study, thermal ablation could be conducted with radiofrequency (RFA) or microwave (MWA).

SUMMARY:
This is a pilot study with a single arm in a single center assessing safety and efficacy of combination therapy of TACE and ablation and durvalumab. This study will be conducted in selected patients with intermediate stage HCC not amenable to curative therapy.

DETAILED DESCRIPTION:
Approximately 30 patients will be enrolled and receive the following treatments:

TACE (day 1, up to twice. TACE interval will be 4～6 weeks) → Ablation (4 weeks after the last TACE, up to twice. Ablation interval will be 4～6 weeks) → Durvalumab (at least 1 week after the last ablation, 1500 mg Q4W, until mRECIST criteria defined radiological progression or other discontinuation criteria were met, but no more than 1 year).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* Age > 18 years.
* Have a HCC diagnosis confirmed by radiology, histology, or cytology. Note: Radiologic confirmation diagnosis is provided by the study site. Definition of radiological confirmation: Clinical findings consistent with the diagnosis of a liver mass measuring at least 1 cm with characteristic vascularization (intense enhancement seen in the hepatic arterial-dominant phase and contrast washout in the late portal venous phase) seen in either triphasic computed tomography (CT) scan or magnetic resonance imaging (MRI).
* HCC newly diagnosed or recurrent with a history of surgery or ablation, with Barcelona Clinic Liver Cancer (BCLC) Stage B not amenable to curative surgery or transplantation or that the patient refuses surgery.
* At least 1 measurable intrahepatic lesion (≥1.0 cm) according to RECISTv1.1 criteria, which is suitable for repeat assessments.
* Tumor size and number requirement: 1 nodule (5cm ≤ size ≤ 7cm); 2-3 nodules, at least 1 nodule > 3cm, and any nodule ≤ 7cm; 4-5 nodules, any nodule size ≤ 7cm;
* Tumors amenable for initial TACE treatment (Permitted modalities are DEB-TACE or cTACE).
* Tumors were assessed with planning ultrasound and suitable for ablation (by experienced doctor to assess and perform ablation procedure).
* Child-Pugh score class A to B7.
* Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Adequate normal organ and marrow function as defined below, Criteria 'a','b','c' and 'f' allow no transfusions, infusions, or growth factor support administered within 14 days before laboratory test: a. Haemoglobin ≤9.0 g/dL; b. Absolute neutrophil count (ANC) ≥1.0 × 10^9 /L; c. Platelet count ≥50 × 10^9/L; d. Serum total bilirubin ≤2 × institutional upper limit of normal (ULN); e. AST (SGOT)/ALT (SGPT) ≤5× ULN; f. Albumin ≥28 g/L; g. International normalized ratio ≤1.6 and prothrombin time ≤16 s; h. Measured creatinine clearance (CL) >50 mL/min or Calculated creatinine CL>50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance: Males: Creatinine CL (mL/min)=Weight (kg) x (140-Age) / (72 x serum creatinine), Females: Creatinine CL (mL/min)=Weight (kg) x (140-Age) ×0.85 / (72 x serum creatinine).
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* History or concurrent use of anticancer therapy (local regional therapy and systemic therapy), including investigational products. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study. Patients with the recurrence from a radical surgery or ablation are allowed. Evidence for radical surgery or ablation should be provided with enhanced MRI/CT after at least 4 weeks after the treatment and AFP level should also be negative in at least 4 weeks after the radical treatment; Chinese traditional medicine with CFDA approval for anticancer use should be washout for 14 days before enrolment.
* Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinoma and HCC, or infiltrative-type HCC
* History of hepatic encephalopathy within past 12 months or requirement for medications to prevent or control encephalopathy
* Ascites requiring invasive intervention (eg, paracentesis) to maintain symptomatic control, within 4 weeks prior to enrolment
* Visible portal vein tumor thrombosis detected on baseline/eligibility imaging
* New York Heart Association Grade ≥2 congestive heart failure; or QTcF value ≥470 ms detected by 12-lead electrocardiogram.
* History of stroke or myocardial infarction or cerebral hemorrhage within 6 months prior to enrolment
* Significant traumatic injury or major surgical procedure (as defined by the Investigator) within 4 weeks prior to enrolment.
* Active GI bleeding, with history of GI bleeding within 6 months, or investigator defined with high risk of haemorrhage for esophageal varices.
* Current use of systemic anticoagulation or anti-platelet drugs.
* History of allogenic organ transplantation.
* Patients weighing ≤30 kg
* Active or prior documented autoimmune or inflammatory disorders. The following are exceptions to this criterion: Patients with vitiligo or alopecia; Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; Any chronic skin condition that does not require systemic therapy; Patients without active disease in the last 5 years may be included; Patients with celiac disease controlled by diet alone
* History of active primary immunodeficiency
* History of another primary malignancy except for: Malignancy treated with curative intent and with no known active disease ≥5 years before the first day of study treatment and of low potential risk for recurrence; Adequately treated non-melanoma skin cancer without evidence of disease; Adequately treated carcinoma in situ without evidence of disease
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice).
* Uncontrolled Hepatitis B (HBV DNA >2000 IU/mL); Patients co-infected with HBV and HCV (characterized by detectable HCV RNA, together with positive HBsAg or detectable HBV DNA according to local laboratory standards). Anti-viral therapy is recommended following the local guidelines. Patients with a non-viral etiology are allowed.
* Current or prior use of immunosuppressive medication within 14 days before enrolment. The following are exceptions to this criterion:a. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection);b. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent;c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication, TACE procedure)
* Uncontrolled intercurrent illness, including but not limited to, unstable angina pectoris, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* History of leptomeningeal carcinomatosis.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Receipt of live attenuated vaccine within 30 days prior to the enrolment. Note: Patients, if enrolled, should not receive live vaccine until 30 days after the last dose of durvalumab.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab.
* Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events | From date of the first treatment until 90 days after the last treatment, assessed up to 21 months
  safety
Serious adverse events | From date of the first treatment until 90 days after the last treatment, assessed up to 21 months
  safety
AEs of Special Interest | From date of the first treatment until 90 days after the last treatment, assessed up to 21 months
  safety
Discontinue rate caused by any AEs | From date of the first treatment until date of the last treatment, assessed up to 18 months
  safety

SECONDARY OUTCOMES:
Progression-free survival (mRECIST) by IRRC | From date of the first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  efficacy
Time to progress (mRECIST) by IRRC | From date of the first treatment until the date of first documented progression, assessed up to 36 months
  efficacy
PFS rate at 12 months (mRECIST) by IRRC | From date of the first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  efficacy
PFS rate at 24 months (mRECIST) by IRRC | From date of the first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  efficacy
Overall survival | From date of the first treatment to the date of death, assessed up to 36 months
  efficacy

IPD SHARING:
Plan to Share IPD: No